CLINICAL TRIAL: NCT07391618
Title: A Study to Evaluate the Efficacy and Safety of a First-line Treatment for Advanced Colorectal Cancer With Simultaneous Infusion of Levozolinate for Injection and 5-FU
Brief Title: Clinical Study on the First-line Treatment of Advanced Colorectal Cancer With Simultaneous Infusion of Levozolinate for Injection and 5-FU
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL-ZY-058
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Advanced Colorectal Cancer
Keywords: levozolinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm1 (Experimental): For patients with wild-type RAS and BRAF and the primary lesion located in the left colorectum, the mFOLFOX6 or FOLFIRI regimens with simultaneous infusion of levofolinic acid and 5-FU for injection were received. Whether to combine cetuximab was determined by the researchers
  Interventions: Drug: mFOLFOX/FOLFIRI ( Standard Chemotherapy)
- arm2 (Experimental): For patients with both RAS and BRAF wild-type and with the primary lesion located in the right colorectal and/or RAS or BRAF mutant type, the mFOLFOX6 or FOLFIRI regimen with simultaneous infusion of levofolinic acid and 5-FU for injection, whether to combine bevacizumab, was determined by the researchers
  Interventions: Drug: mFOLFOX/FOLFIRI ( Standard Chemotherapy)

INTERVENTIONS:
Drug: mFOLFOX/FOLFIRI ( Standard Chemotherapy) — mFOLFOX6: Oxaliplatin 85mg/m², intravenous infusion for 2 hours, day 1; 5-FU 400mg/m² injection, d1; Levofolic acid for injection at 200mg/m² and 5-FU at 2400mg/m² were mixed and infused simultaneously for 46 to 48 hours. Repeat every two weeks until disease progression or intolerable toxicity occurs. FOLFIRI: Irinotecan 180mg/m², intravenous infusion for 30 to 90 minutes on day 1; 5-FU 400mg/m² injection d1; Levofolic acid for injection at 200mg/m² and 5-FU at 2400mg/m² were mixed and infused simultaneously for 46 to 48 hours. Repeat every two weeks until disease progression or intolerable toxicity occurs.

SUMMARY:
Phase II study of simultaneous infusion of levozolinate for injection and 5-FU as first-line treatment for advanced colorectal cancer

DETAILED DESCRIPTION:
To observe and evaluate the efficacy and safety of simultaneous infusion of levofolinate for injection and 5-FU in the first-line treatment of advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined this study and signed the informed consent form.
2. Age: 18 to 75 years old, gender not limited;
3. ECOG PS score: 0-2 points
4. Patients with unresectable or metastatic colorectal cancer confirmed by histology or cytology, where the primary tumor location and the status of RAS and BRAF are known;
5. No previous treatment for unresectable or metastatic lesions has been received;
6. There is at least one measurable lesion in accordance with the RECIST 1.1 standard;
7. In the pre-treatment examination indicators, there was no serious hematopoietic function abnormality, and the functions of the heart, lungs, liver and kidneys were basically normal.

   1. Hemoglobin (Hb) ≥70 g/L;
   2. White blood cell count (WBC) ≥3.0×109/L; Neutrophil count (NEUT) ≥1.5×109/L;
   3. Platelet count (PLT) ≥100×109/L;
   4. Liver function (aspartate aminotransferase AST or alanine aminotransferase ALT) level ≤2.5 times the upper limit of normal value (ULN); Renal function (serum creatinine sCr) level ≤1.5 times the upper limit of the normal value (ULN). Total bilirubin (TBIL) ≤1.5 times the upper limit of the normal value (ULN).
8. The expected survival period is more than three months.

Exclusion Criteria:

1. Those who have been confirmed to be allergic to the test drug and/or its excipients;
2. Those with contraindications to chemotherapy;
3. Colorectal cancer patients with MSI-H or dMMR;
4. Pregnant or lactating women;
5. There is a history of other malignant tumors in the past;
6. Those with systemic internal diseases and mental disorders who are not suitable for chemotherapy;
7. Patients who were determined by the researchers to be unsuitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 3 years

SECONDARY OUTCOMES:
ORR | up to 3 years
DCR | up to 3 years
DoR | up to 3 years
OS | up to 3 years
Adverse Event | Thirty days after the last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Guanghai Dai, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing, China